CLINICAL TRIAL: NCT03658356
Title: Comparison of Verbal Versus Video Instruction in the Collection of Clean Catch Urine in Pregnant Women Undergoing Testing for Asymptomatic Bacturia: Randomized Control Trial
Brief Title: Video Instruction in the Collection of Clean Catch Urine in Pregnant Women Undergoing Testing for Urine Culture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Luke's Hospital, Pennsylvania (Other)
Responsible Party: Principal Investigator, James Anasti, MD, Clinical Professor OB/GYN, St. Luke's Hospital, Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SLIR 2018-89
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Asymptomatic Bacteriuria in Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verbal Instruction on Urine collection (Placebo Comparator): At initial prenatal visit, pregnant patients will be given verbal instructions on how to collect a urinary sample for culture.
  Intervention: Pt will be given verbal instruction to collect urine
  Interventions: Other: Video instructions
- Video instruction on urine collection (Active Comparator): At initial prenatal visit, pregnant patients will watch a video on how to collect a urinary sample for culture
  Intervention: Patient will be asked to watch a video on how to collect a urine sample
  Interventions: Other: Video instructions

INTERVENTIONS:
Other: Video instructions — Pregnant patient will watch her video explaining how to collect a urine sample for asymptomatic bacteriuria determination.

SUMMARY:
The prevalence of asymptomatic bacteriuria in pregnancy has been reported in the range of 2-15%[3]. Due to the severity of the complications related to asymptomatic bacteriuria in this patient population, the American College of OBGYN recommends routine screening of all pregnant women. Asymptomatic bacteriuria in a pregnant woman should be screened only using a clean-catch non contaminated urine sample. Screening for ABU using urine chemistries is not recommended due to the lack of sensitivity and specificity of these tests . If ABU is present, appropriate antibiotic is given and post treatment urine culture is performed. However, a controversy does exist as to the value of treatment of ABU in the prevention of above noted complications [7].

Interestingly, we have noted a contaminated urine cultures in up to 15 to 20% of our prenatal patients. This can be frustrating to both the patient and her physician. Repeat testing, delay in the diagnosis, and additional cost are just some of the problems associated with these contaminated urine cultures.

We hypothesis by improving the instructions given to patients on how to perform a clean catch urine, that we will decease our contaminated urine cultures.

DETAILED DESCRIPTION:
Introduction Asymptomatic bacteriuria (ABU) is defined as the presence of bacteria ( ≥105 per ml) in a non- contaminated urine sample collected from a patient without signs or symptoms related to UTI[1]. Although this is a benign condition that does not require treatment in most adults, ABU in pregnant women has been linked to several complications. The pregnancy state, with its increase in urine stasis and altered immune, can result in increased rates of pyelonephritis and preterm labor[2].

The prevalence of asymptomatic bacteriuria in pregnancy has been reported in the range of 2-15%[3]. Due to the severity of the complications related to asymptomatic bacteriuria in this patient population, the American College of OBGYN recommends routine screening of all pregnant women[4]. Asymptomatic bacteriuria in a pregnant woman should be screened only using a clean-catch non contaminated urine sample. Screening for ABU using urine chemistries is not recommended due to the lack of sensitivity and specificity of these tests[5, 6]. If ABU is present, appropriate antibiotic is given and post treatment urine culture is performed. However, a controversy does exist as to the value of treatment of ABU in the prevention of above noted complications [7].

Interestingly, we have noted a contaminated urine cultures in up to 15 to 20% of our prenatal patients. This can be frustrating to both the patient and her physician. Repeat testing, delay in the diagnosis, and additional cost are just some of the problems associated with these contaminated urine cultures.

Hypothesis/Clinical Question We hypothesis by improving the instructions given to patients on how to perform a clean catch urine, that we will decease our contaminated urine cultures.

Material and Methods:

All patients (16 years and older) presenting for initial routine prenatal care at one of the St Luke University Hospital perinatal clinics will be eligible. Patients with known urinary infection, symptoms of UTI, and other renal disease will be excluded. Consented patients will be randomized (1:1) using previously prepared sealed envelopes to either the current standard of verbal explanation of the clean-catch urine technique or to view the instructional video on the collection technique. A Spanish version video tape will also be available. These sample results as well as basic patient demographics will be collected (Age, Gestational age, BMI, gravidity, parity) will be compared.

We will recruit 200 patients based on an improvement from 15% contaminated rate to a 5% contaminated rate (power 0.80; p=0.05). We will compare proportion of contaminated urine specimens using chi square test to those patients that watch the video to those that did not. In addition, we will compare demographics to determine if any difference exists between the groups. We will employ t-test, chi-squared and Mann-Whitney-U test as appropriate.

Risk and cost to patients This study does not incur any additional risk to the patient. No additional cost will be charged to the patients since all pregnant patients receive a urine culture screen as part of their standard of care.

1. Trautner, B.W., Asymptomatic bacteriuria: when the treatment is worse than the disease. Nat Rev Urol, 2011. 9(2): p. 85-93.
2. Glaser, A.P. and A.J. Schaeffer, Urinary Tract Infection and Bacteriuria in Pregnancy. Urol Clin North Am, 2015. 42(4): p. 547-60.
3. Schneeberger, C., B.M. Kazemier, and S.E. Geerlings, Asymptomatic bacteriuria and urinary tract infections in special patient groups: women with diabetes mellitus and pregnant women. Curr Opin Infect Dis, 2014. 27(1): p. 108-14.
4. Patterson, T.F. and V.T. Andriole, Bacteriuria in pregnancy. Infect Dis Clin North Am, 1987. 1(4): p. 807-22.
5. Rogozinska, E., et al., Accuracy of Onsite Tests to Detect Asymptomatic Bacteriuria in Pregnancy: A Systematic Review and Meta-analysis. Obstet Gynecol, 2016. 128(3): p. 495-503.
6. Awonuga, D.O., et al., Asymptomatic bacteriuria in pregnancy: evaluation of reagent strips in comparison to microbiological culture. Afr J Med Med Sci, 2011. 40(4): p. 377-83.
7. Angelescu, K., et al., Benefits and harms of screening for and treatment of asymptomatic bacteriuria in pregnancy: a systematic review. BMC Pregnancy Childbirth, 2016. 16(1): p. 336.

ELIGIBILITY:
Inclusion Criteria:

* women that are pregnan and requiring a urine sample for asymptomatic bacteriuria testing

Exclusion Criteria:

* any urinary renal disease, including urinary tract infection, proteinuria, hematuria.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09-30 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of contaminated urine specimen | 30 days
  Urines that are contaminated after undergoing culture

IPD SHARING:
Plan to Share IPD: No